CLINICAL TRIAL: NCT03178006
Title: Correlation Between Intestinal Microbiota, Inflamatory Biomarkers, Intestinal Morphology, Hepatic Fibrosis Degree and Vascular Reactivity in Patients With Different Degrees of Glucose Tolerance and Body Adiposity.
Brief Title: Correlation Between Intestinal Microbiota, Inflamatory Biomarkers, Intestinal Morphology, Hepatic Fibrosis Degree and Vascular Reactivity.
Status: Completed | Type: Observational
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Luiz Guilherme Kraemer-Aguiar, MD, Professor, Rio de Janeiro State University
Other Study IDs: 419.676
Record Dates: First submitted 2017-06-03; First posted 2017-06-06 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- healthy controls: healthy individuals
- patients with obesity and dysglycemia: Individuals with BMI > 30 kg/m2 and dysglycemia
- patients with obesity and normoglycemia: Individuals with BMI > 30 kg/m2 and normoglycemia

SUMMARY:
Metabolic, inflammatory status, intestinal permeability biomarkers, and gut microbiota composition were investigated in individuals with varying levels of adiposity and glucose tolerance. This project focuses on exploring the associations between gut permeability and metabolic profiles.

DETAILED DESCRIPTION:
Obese patients with varying levels of adiposity and glucose tolerance from the Obesity Outpatient Clinic, and individuals with normal or overweight weight with dysglycemia or not, preferably from the same social class and type of diet of the obese will be invited to participate in the study. Dysglycemia will be defined by the criteria of the Brazilian Society of Diabetes. These individuals will be divided into three groups: lean controls with normoglycemia (CON), patients with obesity and normoglycemia (NOB), and obesity and dysglycemia (DOB). Biochemical/inflammatory biomarkers, like lipopolysaccharide (LPS) and LPS binding protein (LBP), will be assessed. Duodenal biopsies will be assessed by upper digestive videoendoscopy. Histomorphometry, expression of junctional and cytoskeleton proteins, and enzymatic activity of duodenal epithelium will be used as markers of intestinal permeability. Fecal microbiota composition (FMC) will be analyzed by amplifying the V4 region of the 16S rRNA gene, which will be sequenced with next-generation sequencing technology. Only after approval by the Research Ethics Committee (CEP) of the Pedro Ernesto University Hospital (HUPE-UERJ), will this recruitment begin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women between 18 and 50 years old
* Individuals with obesity and normoglycemia
* Individuals with obesity and dysglycemia

Exclusion Criteria:

* Acute disease
* Chronic pulmonary, cardiovascular, haematological, gastrointestinal, hepatic or renal diseases;
* Unstable dietary history, defined as major changes in diet during the previous month diagnosed by a specialist nutritionist;
* History of gastrointestinal disturbances in activity or chronic diseases, including - inflammatory bowel diseases (IBD), chronic diarrhea of unknown etiology, chronic constipation, disabsorbing syndromes,
* History of major gastrointestinal tract surgery, except cholecystectomy and appendectomy;
* Use of the following medications: probiotics in the last 6 months, systemic antibiotics, oral corticosteroids, cytokines, methotrexate or cytotoxic immunosuppressive agents, consumption of large doses of commercial probiotics (greater than or equal to 10 8 CFU or organisms per day)
* Positive tests for HIV infection and hepatitis B and C;
* Pregnant and lactating women;
* Smokers
* Chronic alcoholism.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese patients with dysglycemia or not from the Obesity Clinic from UERJ will be invited to participate in the study, and individuals with normal or overweight weight with dysglycemia or not, preferably from the same social class and type of diet of the obese
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

PRIMARY OUTCOMES:
Correlation | 2018
  We hypothesize that greater glucose intolerance and obesity are associated with higher epithelial barrier dysfunction and changes in fecal microbiota composition (FMC). We investigated the metabolic and inflammatory biomarkers, intestinal permeability, and FMC in normoglycemic controls versus normoglycemic and dysglycemic individuals with obesity. Specifically, we tested the associations between intestinal permeability and metabolic markers.

IPD SHARING:
Plan to Share IPD: No